CLINICAL TRIAL: NCT03626766
Title: A Randomized Controlled Trial Evaluating the Effectiveness of Displaying Patient Photographs in an Electronic Health Record to Prevent Wrong-Patient Electronic Orders
Brief Title: Evaluating the Impact of Patient Photographs for Preventing Wrong-Patient Errors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Montefiore Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAR0080; R01HS024713 (AHRQ); R01HD094793 (NIH)
Record Dates: First submitted 2018-08-06; First posted 2018-08-13 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Medical Errors; Electronic Medical Records
Keywords: Allscripts; Epic; Electronic Health Record (EHR); Electronic orders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Photo in Verification Alert (Active Comparator): Patient photo displayed in a patient ID verification alert when placing electronic orders in the electronic health record.
  Interventions: Behavioral: Photo in Verification Alert
- Photo in Banner (Active Comparator): Patient photo displayed in the banner (at the top of the screen).
  Interventions: Behavioral: Photo in Banner
- Photo in Banner and Verification Alert (Active Comparator): Patient photograph displayed in the banner (at the top of the screen) AND patient photo displayed in a verification alert when placing electronic orders.
  Interventions: Behavioral: Photo in Banner and Verification Alert
- No Photo (No Intervention): No patient photographs displayed in the electronic health record.

INTERVENTIONS:
Behavioral: Photo in Verification Alert — Patient photograph displayed in a patient ID verification alert when placing electronic orders in the electronic health record.
  Arms: Photo in Verification Alert
Behavioral: Photo in Banner — Patient photograph will be displayed in the banner at the top of the screen in the electronic health record.
  Arms: Photo in Banner
Behavioral: Photo in Banner and Verification Alert — Patient photograph will be displayed in the banner at the top of the screen in the electronic health record AND patient photograph displayed in a patient ID verification alert when placing electronic orders in the electronic health record.
  Arms: Photo in Banner and Verification Alert

SUMMARY:
This is a multi-site, 4-arm randomized controlled trial to test the effectiveness of patient photographs displayed in electronic health record (EHR) systems to prevent wrong-patient order errors. The study will be conducted at several academic medical centers that utilize two different EHR systems. Because EHR systems have different functionality for displaying patient photographs, two different study designs will be employed. In Allscripts EHR, a 2-arm randomized trial will be conducted in which providers are randomized to view order verification alerts with versus without patient photographs when placing electronic orders. In Epic EHR, a 2x2 factorial trial will be conducted in which providers are randomized to one of four conditions: 1) no photograph; 2) photograph displayed in the banner only; 3) photograph displayed in a verification alert only; or 4) photograph displayed in the banner and verification alert. The main hypothesis of this study is that displaying patient photographs in the EHR will significantly reduce the frequency of wrong-patient order errors, providing health systems with the evidence needed to adopt this safety practice.

DETAILED DESCRIPTION:
Although Computerized provider order entry (CPOE) systems are associated with a reduction in medical errors, when orders are placed electronically certain types of errors, including placing orders on the wrong patient, may occur more frequently. The danger of wrong-patient electronic orders was highlighted by one hospital's report of over 5,000 wrong patient orders in 1 year. With the growing use of electronic health records (EHRs), an effective method to minimize wrong-patient orders is needed. One study showed that patient photographs displayed in EHR systems decreased wrong-patient orders from 12 to 3 per year after patient photographs were implemented. While encouraging, this study was limited due to its small sample size, compared outcomes of the intervention participants to outcomes of a comparison group similar in demographics but may have differed in ways that were not measured in the study (quasi-experimental design), and reliance on voluntary reporting of errors by providers, which is known to be unreliable and greatly underestimate the actual error rate. This research proposes to use an automated and reliable measure of wrong-patient errors instead of voluntary reporting will demonstrate that patient photographs can significantly prevent wrong-patient orders.

ELIGIBILITY:
Inclusion Criteria:

* All patients for whom an order was placed in the study period.
* All providers with the authority to place electronic orders and who placed electronic orders during the study period.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10426 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason S. Adelman, MD, MS, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York
  - Weill Cornell Medical Center - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adelman JS, Kalkut GE, Schechter CB, Weiss JM, Berger MA, Reissman SH, Cohen HW, Lorenzen SJ, Burack DA, Southern WN. Understanding and preventing wrong-patient electronic orders: a randomized controlled trial. J Am Med Inform Assoc. 2013 Mar-Apr;20(2):305-10. doi: 10.1136/amiajnl-2012-001055. Epub 2012 Jun 29. PMID 22753810

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Photo in Verification Alert | Photo in Banner | Photo in Banner and Verification Alert | No Photo
Started | 2610 | 2608 | 2602 | 2606
Completed | 2171 | 2202 | 2196 | 2199
Not Completed | 439 | 406 | 406 | 407

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Photo in Verification Alert | Photo in Banner | Photo in Banner and Verification Alert | No Photo | Total
Number analyzed (Participants) | 2171 | 2202 | 2196 | 2199 | 8768
Age, Customized [Count of Participants; unit: Participants]
  >18 years | 2171 | 2202 | 2196 | 2199 | 8768
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex and gender were not collected from any participant.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2171 | 2202 | 2196 | 2199 | 8768

OUTCOME MEASURES:

1. Primary Outcome: Number of Order Sessions With at Least One Retract-and-Reorder (RAR) Event as Identified by the Wrong-Patient Retract-and-Reorder (RAR) Measure.
Description: Using the Wrong-Patient (WP) Retract-and-Reorder measure, the outcome was WP order sessions, defined as series of orders placed by 1 clinician for 1 patient that included ≥1 WP order. The Wrong-Patient Retract-and-Reorder (RAR) measure is an automated, validated, and reliable measure endorsed by the National Quality Forum (NQF #2723). The RAR measure identifies orders placed for a patient that are retracted within 10 minutes, and then placed by the same provider for a different patient within the next 10 minutes. These are near-miss errors, self-caught by the provider before they reach the patient and cause harm.
Time Frame: 2 years
Measure: Number; unit: WP Order Sessions
Units Other Than Participants: order sessions
Arm/Group | Photo in Verification Alert | Photo in Banner | Photo in Banner and Verification Alert | No Photo
Number analyzed (Participants) | 2171 | 2202 | 2196 | 2199
Number analyzed (order sessions) | 3948077 | 3958269 | 4028011 | 4007833
WP Order Sessions | 5587 | 5836 | 5598 | 6279

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 2 years (11/17/2021 - 11/16/2023).
Arm/Group | Photo in Verification Alert | Photo in Banner | Photo in Banner and Verification Alert | No Photo
All-Cause Mortality (participants affected / at risk) | 0/2171 | 0/2202 | 0/2196 | 0/2199
Serious Adverse Events (participants affected / at risk) | 0/2171 | 0/2202 | 0/2196 | 0/2199
Other Adverse Events (participants affected / at risk) | 0/2171 | 0/2202 | 0/2196 | 0/2199

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03626766/Prot_SAP_000.pdf